CLINICAL TRIAL: NCT04371211
Title: Telemedicine Brain Injury Coping Skills (BICS-T) Support Group for Brain Injury Survivors and Their Caregivers: A Feasibility Study
Brief Title: Telemedicine Brain Injury Coping Skills (BICS-T) Support Group for Brain Injury Survivors and Their Caregivers
Acronym: BICS-T I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rehabilitation Hospital of Indiana (Other)
Responsible Party: Principal Investigator, Devan Parrott, Director and Biostatistician, Rehabilitation Hospital of Indiana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1808716960
Record Dates: First submitted 2019-08-07; First posted 2020-05-01 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Traumatic Brain Injury; Coping Skills
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Feasibility Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Telemedicine Brain Injury Coping Skills — BICS is a 12 session (one session per week), manualized, cognitive-behavioral treatment group designed to provide support, coping skills, and psychoeducation aimed to improve perceived self-efficacy (PSE) and emotional functioning. PSE has been found to be strongly linked to social participation, increased positive regard toward the caregiving role, and was found to be the greatest contributing factor to predicting life satisfaction.
  For this study, the Brain Injury Coping Skills (BICS) group intervention will be administered electronically in a web-based group telemedicine platform, BICS-T. The purpose of this phase is to test the feasibility, participant training protocol, and ease of use of equipment and technology.

SUMMARY:
Brain Injury can be devastating for both patients and family members and can result in chronic difficulties in vocational, social, financial, as well as physical functioning. The occurrence of emotional and neurobehavioral challenges in individuals with brain injury is also common with research consistently showing links between these challenges and a person's overall rehabilitation outcome. In order to provide patients and caregivers greater support and teach adaptive coping strategies, the authors of this grant designed and studied a coping skills group specifically for brain injury survivors and their caregivers at the Rehabilitation Hospital of Indiana (RHI) called the Brain Injury Coping Skills group (BICS). BICS is a 12 session (one session per week), manualized, cognitive-behavioral treatment group designed to provide support, coping skills, and psychoeducation aimed to improve perceived self-efficacy (PSE) and emotional functioning.

DETAILED DESCRIPTION:
Brain Injury can be devastating for both patients and family members and can result in chronic difficulties in vocational, social, financial, as well as physical functioning.The occurrence of emotional and neurobehavioral challenges in individuals with brain injury is also common with research consistently showing links between these challenges and a person's overall rehabilitation outcome. Additionally, family functioning and caregiver well-being has been shown to influence rehabilitation outcome for a survivor after brain injury.In fact, individuals with families and caregivers who receive support and services, as well as learn adaptive coping strategies, are less likely to exhibit these marked levels of psychological distress.

In order to provide patients and caregivers greater support and teach adaptive coping strategies, the authors of this grant designed and studied a coping skills group specifically for brain injury survivors and their caregivers at the Rehabilitation Hospital of Indiana (RHI) called the Brain Injury Coping Skills group (BICS). BICS is a 12 session (one session per week), manualized, cognitive-behavioral treatment group designed to provide support, coping skills, and psychoeducation aimed to improve perceived self-efficacy (PSE) and emotional functioning. Perceived self-efficacy is the belief or confidence in one's ability to deal with the challenges related to a specific situation (e.g., brain injury). PSE has been found to be strongly linked to social participation, increased positive regard toward the caregiving role, and was found to be the greatest contributing factor to predicting life satisfaction. Cicerone and Azulay found that the greatest contribution to predicting life satisfaction was the person's PSE for managing their cognitive challenges.

Fourteen participants will be recruited. Participants with brain injury or caregivers of brain injury survivors who meet inclusion/exclusion criteria will be recruited by the research associate. At baseline, participants will be asked to come to the Rehabilitation Hospital of Indiana's Neuro Rehabilitation Center (RHI NRC) to collect study equipment and complete baseline data collection. First, participants will be provided an IPad and training on using the IPad and study software. Specifically, participants will be trained on turning on the IPad, finding the app for the study groups, signing into the app, and using the app to participate in the group sessions. A simulation session will also be provided to ensure participants can login, access the software, and interact during a session. After training, participants will be provided take home instructions and contact information for the research assistant for at home troubleshooting if needed. Also after training, the research assistant will ask participants to provide feedback on the training. The research assistant will also ask participants to complete some questionnaires during this visit including a survey including demographics as well as primary and secondary outcome measures. The visit is expected to take between one and two hours and this portion of the study will be completed face to face. Participants will then be asked to participate in BICS-T. BICS-T is a group intervention that will take place over telemedicine software on the IPad provided to participants. Sessions will occur once a week for 12 weeks. Each session will last two hours. This portion of the study is completed 100% on the IPad and will not require any transportation to NRC. After BICS-T is over (after all 12 sessions = 12 weeks), participants will be asked to return to RHI NRC to complete post-test surveys and return the equipment that participants receive after participants have completed the program. This final session is expected to take approximately two hours.

ELIGIBILITY:
Inclusion Criteria:

* Persons with a history of brain injury (e.g., Traumatic Brain Injury; TBI) or acquired BI such as stroke, hypoxia, ruptured aneurysm, or metabolic encephalopathy);
* 18 years of age and older;
* at least six months post-injury; and
* able to speak English fluently.

Exclusion Criteria:

* at imminent risk of psychiatric breakdown, or in imminent danger of hurting themselves or others;
* active psychosis;
* aphasia that limits group participation;
* significant neurobehavioral difficulties that would be deemed disruptive to group participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Brain Injury Self-Efficacy Scale | Through study completion, up to 5 months
  Assesses perceived self-efficacy regarding a person's brain injury and proved responsive to treatment effects in the original BICS study. Participants identify how confident they are about various statements from 0 (Not at all) to 4 (Extremely). Item scores are totaled and higher scores suggest higher reported self-efficacy.

SECONDARY OUTCOMES:
The Group Climate Questionnaire | Through study completion, up to 5 months
  This measure is the most commonly used group process instrument. It is a self-report, 12-item questionnaire that assesses the person's perceptions of the group's therapeutic environment. Items are scored on a 7-point Likert scale ranging from "Not at all" to "Extremely." The three subscales includes Engagement (the level of positive working group atmosphere), Conflict (the level of anger and tension in the group), and Avoidance (the level of behaviors indicating avoidance of personal responsibility of group work by the members). Higher scores are linked with greater perceived group cohesiveness and positive environment.
The Client Satisfaction Questionnaire | Through study completion, up to 5 months
  This measure determines perceived satisfaction with the program (e.g., To what extent has the investigator's program met your needs?) Have the services you received helped you to deal more effectively with your problems?) Scores range from 8-32 (higher scores indicate higher satisfaction).
Patient-reported outcome measurement information system (PROMIS): Self-efficacy for managing symptoms | Through study completion, up to 5 months
  This measures a person's confidence in managing one's daily activities, emotions, medications/treatments, social interactions, and symptoms. Participants rate their level of confidence for various items on a scale of 1 (I am not at all confident) to 5 (I am very confident). Higher scores suggest greater self-efficacy.
Quality of life after brain injury: scale | Through study completion, up to 5 months
  This is a quality of life measure designed specifically for patients with brain injury. It measures patient's reported quality of life after their brain injury. Participants respond to items, indicating how satisfied they are with the items, using a scale from 1 (Not at all) to 5 (Very). Item scores are added up. Higher scores suggest greater quality of life.
Patient-reported outcome measurement information system (PROMIS): Health-related quality of life | Through study completion, up to 5 months
  This is an evaluation of a person's overall quality of life based on physical limitations and ability to participate socially. Participants respond to various items using a scale of 1 (I am not at all confident) to 5 (I am very confident). Higher scores suggest greater quality of life.
Therapeutic Factors Inventory | Through study completion, up to 5 months
  This measures one's feeling of acceptance in a group setting, as well as sense of belonging, working together, trust, and caring. Participants respond to various items using a scale of 1 (Strongly disagree) to 7 (Strongly agree). Greater scores suggest greater feelings of support and group cohesion.
Technology and Internet Assessment | Through study completion, up to 5 months
  This is an assessment that evaluates a participant's strengths and weaknesses in understanding computers, the Internet, and information technology skills. Higher scores indicate greater use of and skills with the internet and technology.

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Hospital of Indiana, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No